CLINICAL TRIAL: NCT05517603
Title: A Phase 1/2a, Randomized, Double-Blind, Placebo-Controlled, First-In-Patient Study Of AJ201 To Evaluate Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics In Adults With Spinal And Bulbar Muscular Atrophy (SBMA)
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Of AJ201 In Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AnnJi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JM17-201-201
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-05

CONDITIONS: Spinal and Bulbar Muscular Atrophy; Kennedy's Disease
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: AJ201 (Active Comparator): Subjects taking active drug AJ201 600mg/day for 12 weeks.
  Interventions: Drug: AJ201
- Placebo Comparator (Placebo Comparator): Subjects taking placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AJ201 — Administered orally
  Other Names: JM17
  Arms: Experimental: AJ201
Drug: Placebo — Administered orally
  Arms: Placebo Comparator

SUMMARY:
This is a phase 1/2a randomized, double-blind study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of study drug AJ201 in subjects with Spinal and Bulbar Muscular Atrophy (SBMA).

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent before any assessment is performed.
2. Adult males aged 18 or greater with a confirmed genetic diagnosis (confirmed CAG repeat expansion in the AR gene of at least 36 repeat) of SBMA and clinical diagnosis of symptomatic muscle weakness.
3. Able to complete 2MWT with or without the aid of an assisted device at screening.
4. SBMAFRS score ≥26 (subjects with moderate to high physical performance) at screening.
5. Willing to participate in all aspects of study design and assessments, including blood draw and muscle biopsies.
6. Male subjects and their female spouses/partners who are of childbearing potential must agree to use highly effective contraception consisting of 2 forms of birth control (at least 1 of which must be a barrier method) starting from the first dose of the study drug and continuing throughout the study period and for 90 days after the last dose of the study drug. Male subjects should also not donate sperm during the study and for 90 days after the final administration of the study drug.
7. Able to communicate well with the Investigator, to understand, and comply with the requirements of the study.

Exclusion Criteria:

1. Nonambulatory.
2. Contraindications to MRI such as a contraindicated nonremovable metal device (ie, pacemaker, defibrillator, insulin pump, metal clips, nonremovable jewelry) or claustrophobia.
3. Use of other investigational products within 30 days, or within 5 half-lives, whichever is longer, prior to the first dosing, or until the expected PD effect has returned to baseline, whichever is longer. Approved COVID-19 vaccines are not considered investigational treatments and are allowed prior to, during, and after the study.
4. Use of drugs known to affect muscle metabolism within the previous 1 month prior to the first dosing, including (but not limited to) systemic corticosteroids (>10 mg/day prednisone or equivalent), androgens, or androgen reducing agents, systemic beta agonists or beta blockers, and relevant herbal, or nutraceutical products. For subjects using systemic corticosteroids (≤10 mg/day or equivalent), they should be on stable dose for the previous 3 months prior to first dosing.
5. Known history of allergic reactions to curcumin analogs or excipients in the study drug formulation.
6. Known history of clinically significant cardiovascular disease (including uncontrolled hypertension, ischemic heart disease [eg, myocardial infarction, angina, abnormal coronary arteriography or cardiac stress testing/imaging]), heart failure or left ventricle dysfunction of New York Heart Association Classification III-IV, or clinically significant cerebrovascular disease (stroke or transient ischemic attacks).
7. An abnormal ECG at screening visit which is judged to be clinically relevant and represents an unacceptable risk for study participation by the Investigator. An example is Brugada-like ECG changes which have been reported in SBMA patients in Italy and Japan.
8. Any surgical or medical condition which may jeopardize the subject in case of participation in the study. The Investigator should make this determination in consideration of the subject's medical history and/or clinical or laboratory evidence of any of the following during screening:

   1. Liver disease or liver injury as indicated by abnormal liver function tests such as AST, ALT, gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP), or serum bilirubin in the presence of normal serum creatine kinase (CK).
   2. Significant swallowing dysfunction, which may increase the risk of accidental choking and aspiration pneumonia.
9. Subjects with renal impairment defined as a creatinine clearance of <90 mL/min at screening. (Creatinine Clearance = [140 - age in years] *weight in kg]/[72*serum Cr(mg/dL)]).
10. History of active tuberculosis or exposure to endemic areas within 8 weeks prior to QuantiFERON®-TB testing performed at screening.
11. Positive QuantiFERON®-TB indicating possible tuberculosis infection.
12. History of immunodeficiency diseases, including a positive HIV test result at screening.
13. A positive hepatitis B surface antigen or hepatitis C test result at screening.
14. Subjects with known bleeding disorders, or who are under treatment with anticoagulants or with a platelet count <50,000 (due to the increased risk of bleeding during muscle biopsy procedure).
15. History of drug or alcohol abuse within the 12 months prior to the first dosing, or evidence of such abuse as indicated by the laboratory assays conducted during screening.
16. The Investigator should be guided by the following criteria during screening: a. Any single laboratory parameter may not exceed 3 times the upper limit of normal (ULN). A single parameter elevated up to and including 3 times the ULN should be re-checked once more as soon as possible, and in all cases, at least prior to enrollment/randomization, to rule out lab error. For abnormal liver function tests, in the presence of elevated serum CK levels, ALT, or AST, up to 5 times the ULN are acceptable if other liver tests are normal. b. If the total bilirubin concentration is increased above 1.5 times the ULN, total bilirubin should be differentiated into the direct and indirect reacting bilirubin. In any case, serum indirect bilirubin should not exceed the value of 1.6 mg/dL (27 mol/L).
17. Use of drugs that are inhibitors of CYP3A4, 2B6, or 2C19 within 2 weeks prior to the first dosing and during the study.
18. Use of drugs that are substrates of MATE1 or MATE2-K transporters within 2 weeks prior to the first dosing and during the study.
19. Use of turmeric or products containing curcumin within 2 weeks prior to the first dosing and during the study.
20. Use of aspirin or nonsteroidal anti-inflammatory agents within 3 days prior to the baseline visit (due to the increased risk of bleeding during muscle biopsy procedure).
21. Any reason that, in the opinion of the Investigator, would prevent the subject from participating in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Incidence and proportion of subjects with AEs including SAEs and TEAEs. | 12 weeks
  Safety will be monitored throughout the study.

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Plasma Concentration (Cmax) will be assessed | Visit 3/Week 2 and Visit 4/Week 6 at the following time points: predose and 0.5, 1, 2, 4, 8, and 12 hours postdose.
  Blood sampling will be collected at Visit 3 and Visit 4.
Pharmacokinetics: Area Under the Curve (AUC) will be assessed | Visit 3/Week 2 and Visit 4/Week 6 at the following time points: predose and 0.5, 1, 2, 4, 8, and 12 hours postdose.
  Blood sampling will be collected at Visit 3 and Visit 4.
Pharmacodynamics: Change from baseline in mutant androgen receptor protein levels in skeletal muscle in treatment vs placebo group. | Visit 2/Week 1 and Visit 5/Week 12
  Samples will be collected at Visit 2 and Visit 5.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California, Irvine, Orange, California
  - Stanford University, Palo Alto, California
  - Mayo Clinic, Jacksonville, Florida
  - National Institutes of Health, Bethesda, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No